CLINICAL TRIAL: NCT02985957
Title: A Phase 2 Trial of Nivolumab Plus Ipilimumab, Ipilimumab Alone, or Cabazitaxel in Men With Metastatic Castration-Resistant Prostate Cancer
Brief Title: A Study of Nivolumab Plus Ipilimumab, Ipilimumab Alone, or Cabazitaxel in Men With Metastatic Castration-Resistant Prostate Cancer (CheckMate 650)
Acronym: CheckMate 650
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-650; 2016-001928-54 (EudraCT Number)
Record Dates: First submitted 2016-11-22; First posted 2016-12-07 (Estimated); Results first posted 2023-04-24 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Nivolumab; Ipilimumab; cabazitaxel; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Cohort A (Arm A) (Experimental)
  Interventions: Biological: Nivolumab; Biological: Ipilimumab
- Cohort B (Arm B) (Experimental)
  Interventions: Biological: Nivolumab; Biological: Ipilimumab
- Cohort C (Arm C) (Experimental)
  Interventions: Biological: Nivolumab; Biological: Ipilimumab
- Cohort D (Arm D1) (Experimental)
  Interventions: Biological: Nivolumab; Biological: Ipilimumab
- Cohort D (Arm D2) (Experimental)
  Interventions: Biological: Nivolumab; Biological: Ipilimumab
- Cohort D (Arm D3) (Experimental)
  Interventions: Biological: Ipilimumab
- Cohort D (Arm D4) (Experimental)
  Interventions: Drug: Cabazitaxel; Drug: Prednisone

INTERVENTIONS:
Biological: Nivolumab — Specified dose on specified days
  Other Names: BMS-936558; Opdivo
  Arms: Cohort A (Arm A); Cohort B (Arm B); Cohort C (Arm C); Cohort D (Arm D1); Cohort D (Arm D2)
Biological: Ipilimumab — Specified dose on specified days
  Other Names: BMS-734016; Yervoy
  Arms: Cohort A (Arm A); Cohort B (Arm B); Cohort C (Arm C); Cohort D (Arm D1); Cohort D (Arm D2); Cohort D (Arm D3)
Drug: Cabazitaxel — Specified dose on specified days
  Arms: Cohort D (Arm D4)
Drug: Prednisone — Specified dose on specified days
  Arms: Cohort D (Arm D4)

SUMMARY:
The purpose of this study is to evaluate the effectiveness, safety and tolerability of nivolumab followed by ipilimumab, in subjects with metastatic castration resistant prostate cancer (mCRPC).

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Current evidence of metastatic disease documented by either bone lesions on radionuclide bone scan and/or soft tissue lesions on computerized tomography/magnetic resonance imaging (CT/MRI).
* Ongoing androgen deprivation therapy (ADT) with a Gonadotropin-releasing hormone (GnRH) analogue or a surgical/medical castration with testosterone level of ≤1.73nmol/L (50ng/dL)

For crossover phase for participants originally randomized to Arm D3 or Arm D4 only:

* Previously randomized to Arm D3 or D4; had histologic confirmation of adenocarcinoma of the prostate and evidence of Stage IV disease (as defined by American Joint Committee of Cancer criteria (AJCC criteria) prior to randomization

Exclusion Criteria:

* Presence of visceral metastases in the liver
* Active brain metastases or leptomeningeal metastases
* Active, known, or suspected autoimmune disease or infection
* Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, or anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways

For crossover phase for participants originally randomized to Arm D3 or Arm D4 only:

* Prior radiation therapy within 14 days prior to first dose of nivolumab combined with ipilimumab
* Have received systemic anti-cancer therapy after the last dose of study treatment (ipilimumab or cabazitaxel)

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 351 (Actual)
Dates: Start 2017-03-26 (Actual); Primary Completion 2022-04-05 (Actual); Study Completion 2025-01-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (59):
- United States (15):
  - Local Institution - 0074, Tucson, Arizona
  - Local Institution - 0046, Marietta, Georgia
  - Local Institution - 0011, Chicago, Illinois
  - Local Institution - 0076, Minneapolis, Minnesota
  - Local Institution - 0008, St Louis, Missouri
  - Local Institution - 0075, Las Vegas, Nevada
  - Local Institution - 0078, Albany, New York
  - Local Institution - 0065, Lake Success, New York
  - Local Institution - 0001, New York, New York
  - Local Institution - 0077, Tigard, Oregon
  - Local Institution - 0047, Allentown, Pennsylvania
  - Local Institution - 0010, Philadelphia, Pennsylvania
  - Local Institution - 0067, Charleston, South Carolina
  - Local Institution - 0079, Austin, Texas
  - Local Institution - 0002, Houston, Texas
- Australia (7):
  - Local Institution - 0027, Gosford, New South Wales
  - Local Institution - 0059, Wahroonga, New South Wales
  - Local Institution - 0029, Westmead, New South Wales
  - Local Institution - 0028, Southport, Queensland
  - Local Institution - 0043, Woolloongabba, Queensland
  - Local Institution - 0030, Elizabeth Vale, South Australia
  - Local Institution - 0031, Clayton, Victoria
- Local Institution - 0048, Vienna, Austria
- Local Institution - 0044, Montreal, Quebec, Canada
- Denmark (4):
  - Local Institution - 0063, Aarhus N, Central Jutland
  - Local Institution - 0062, Aalborg
  - Local Institution - 0061, København Ø
  - Local Institution - 0060, Odense
- France (4):
  - Local Institution - 0009, Clermont-Ferrand
  - Local Institution - 0005, Lyon
  - Local Institution - 0004, Marseille
  - Local Institution - 0003, Villejuif
- Germany (12):
  - Local Institution - 0038, Göttingen, Lower Saxony
  - Local Institution - 0041, Braunschweig
  - Local Institution - 0032, Dresden
  - Local Institution - 0019, Herne
  - Local Institution - 0017, Jena
  - Local Institution - 0034, Munich
  - Local Institution - 0018, Münster
  - Local Institution - 0037, Nuremberg
  - Local Institution - 0042, Nürtingen
  - Local Institution - 0036, Rostock
  - Local Institution - 0033, Tübingen
  - Local Institution - 0035, Wesel
- Italy (5):
  - Local Institution - 0071, Arezzo
  - Local Institution - 0052, Milan
  - Local Institution - 0053, Napoli
  - Local Institution - 0072, Parma
  - Local Institution - 0051, Terni
- Poland (3):
  - Local Institution - 0055, Krakow, Lesser Poland Voivodeship
  - Local Institution - 0066, Koszalin
  - Local Institution - 0054, Warsaw
- Spain (7):
  - Local Institution - 0022, Madrid, Sede Madrid
  - Local Institution - 0026, Badajoz
  - Local Institution - 0025, Barcelona
  - Local Institution - 0020, Madrid
  - Local Institution - 0021, Madrid
  - Local Institution - 0024, Málaga
  - Local Institution - 0023, Santiago Compostela

REFERENCES:
- [Derived] Sharma P, Pachynski RK, Narayan V, Flechon A, Gravis G, Galsky MD, Mahammedi H, Patnaik A, Subudhi SK, Ciprotti M, Simsek B, Saci A, Hu Y, Han GC, Fizazi K. Nivolumab Plus Ipilimumab for Metastatic Castration-Resistant Prostate Cancer: Preliminary Analysis of Patients in the CheckMate 650 Trial. Cancer Cell. 2020 Oct 12;38(4):489-499.e3. doi: 10.1016/j.ccell.2020.08.007. Epub 2020 Sep 10. PMID 32916128
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Cohort A: Asymptomatic or minimally symptomatic, not previously received second generation hormone therapies or cytotoxic chemotherapy.
  Cohort B: Asymptomatic or minimally symptomatic, progressed after second generation hormone therapies and had not been treated with cytotoxic chemotherapy.
  Cohort C: Progressed after prior taxane-based cytotoxic chemotherapy. Cohort D: Progressed after prior docetaxel-containing therapy.
Groups:
- Cohort A: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg: Part 1: Nivolumab 1 mg/kg as a 30-minute IV infusion, on Day 1 of each treatment cycle every 3 weeks for 4 doses (Cycles 1-4), then ipilimumab 3 mg/kg as a 30-minute IV infusion, on Day 1 of each treatment cycle every 3 weeks for 4 doses (Cycles 1-4). Part 2: Not reached for this cohort - Six weeks after the last co-administered dose in Part 1, a flat dose of 480 mg nivolumab on Day 1 of each 4-week treatment cycle given IV given over approximately 30 minutes every 4 weeks until unacceptable toxicity or disease progression.
- Cohort B: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg; Cohort C: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg: Part 1: Nivolumab 1 mg/kg as a 30-minute IV infusion, on Day 1 of each treatment cycle every 3 weeks for 4 doses (Cycles 1-4), then ipilimumab 3 mg/kg as a 30-minute IV infusion, on Day 1 of each treatment cycle every 3 weeks for 4 doses (Cycles 1-4). Part 2: Six weeks after the last co-administered dose in Part 1, a flat dose of 480 mg nivolumab on Day 1 of each 4-week treatment cycle given IV given over approximately 30 minutes every 4 weeks until unacceptable toxicity or disease progression.
- Cohort D Arm 1: Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg Q3W: Nivolumab 3 mg/kg in combination with ipilimumab 1 mg/kg every 3 weeks for up to 4 doses (Cycles 1 to 4), followed by nivolumab 480 mg administered every 4 weeks (Cycle 5 and beyond). Participants receiving maintenance nivolumab with ongoing disease control or with radiographic progression were permitted re-induction with the combination of ipilimumab and nivolumab at their original combination dose upon PSA progression or radiographic progression (whichever occured first). Treatment continued until disease progression, unacceptable toxicity, withdrawal of consent, 2-year maximum treatment duration, or the study ends, whichever occurred first.
- Cohort D Arm 2: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg Q6W: Nivolumab 1 mg/kg every 3 weeks plus ipilimumab 3 mg/kg every 2 cycles (ie, every 6 weeks) for up to 4 ipilimumab doses, followed by nivolumab 480 mg every 4 weeks. Participants receiving maintenance nivolumab with ongoing disease control or with radiographic progression were permitted reinduction with the combination of ipilimumab and nivolumab at their original combination dose upon PSA progression or radiographic progression (whichever occurred first). Treatment continued until disease progression, unacceptable toxicity, withdrawal of consent, 2-year maximum treatment duration, or the study ended, whichever occurred first.
- Cohort D Arm 3: Ipilimumab 3 mg/kg: Ipilimumab 3 mg/kg every 3 weeks for up to 4 doses. Treatment continued until disease progression, unacceptable toxicity, withdrawal of consent, completion of 4 cycles, or the study ended, whichever occurred first. Participants who progressed on or after treatment were eligible to crossover to Arm D1.
- Cohort D Arm 4: Cabazitaxel 20 mg/m2 or 25 mg/m2 + Prednisone 10 mg: Cabazitaxel 20 mg/m2 or 25 mg/m2 (at investigator's discretion and according to country-specific label) every 3 weeks in combination with oral prednisone or prednisolone 10 mg daily for up to 10 cycles. Treatment continued until disease progression, unacceptable toxicity, withdrawal of consent, completion of 10 cycles of treatment, or the study ended, whichever occurred first. Participants who progressed on or after treatment were eligible to crossover to Arm D1.
Period: Pre-Treatment Period
Arm/Group | Cohort A: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg | Cohort B: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg | Cohort C: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg | Cohort D Arm 1: Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg Q3W | Cohort D Arm 2: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg Q6W | Cohort D Arm 3: Ipilimumab 3 mg/kg | Cohort D Arm 4: Cabazitaxel 20 mg/m2 or 25 mg/m2 + Prednisone 10 mg
Started | 2 | 45 | 45 | 73 | 74 | 38 | 74
Completed | 2 | 45 | 45 | 73 | 73 | 38 | 72
Not Completed | 0 | 0 | 0 | 0 | 1 | 0 | 2
Not completed — Participant no longer meets study criteria | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Participant withdrew consent | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Adverse event unrelated to study drug | 0 | 0 | 0 | 0 | 0 | 0 | 1
Period: Treatment Period
Arm/Group | Cohort A: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg | Cohort B: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg | Cohort C: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg | Cohort D Arm 1: Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg Q3W | Cohort D Arm 2: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg Q6W | Cohort D Arm 3: Ipilimumab 3 mg/kg | Cohort D Arm 4: Cabazitaxel 20 mg/m2 or 25 mg/m2 + Prednisone 10 mg
Started (Started Treatment) | 2 | 45 | 45 | 73 | 73 | 38 | 72
Eligible Participants Who Progressed and Received Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg | 0 | 0 | 0 | 0 | 0 | 13 | 27
Completed | 0 | 0 | 0 | 5 | 3 | 19 | 25
Not Completed | 2 | 45 | 45 | 68 | 70 | 19 | 47
Not completed — Death | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Participant withdrew consent | 0 | 0 | 0 | 1 | 3 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Other reasons | 0 | 0 | 1 | 3 | 5 | 0 | 1
Not completed — Not reported | 0 | 2 | 2 | 5 | 0 | 0 | 0
Not completed — Maximum clinical benefit | 0 | 0 | 1 | 1 | 0 | 0 | 2
Not completed — Adverse event unrelated to study drug | 1 | 4 | 1 | 2 | 8 | 2 | 7
Not completed — Study drug toxicity | 1 | 23 | 20 | 12 | 20 | 3 | 5
Not completed — Disease progression | 0 | 16 | 20 | 40 | 29 | 11 | 28
Not completed — Participant request to discontinue study treatment | 0 | 0 | 0 | 4 | 2 | 2 | 3
Not completed — Poor/Non-Compliance | 0 | 0 | 0 | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg | Cohort B: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg | Cohort C: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg | Cohort D Arm 1: Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg Q3W | Cohort D Arm 2: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg Q6W | Cohort D Arm 3: Ipilimumab 3 mg/kg | Cohort D Arm 4: Cabazitaxel 20 mg/m2 or 25 mg/m2 + Prednisone 10 mg | Total
Number analyzed (Participants) | 2 | 45 | 45 | 73 | 74 | 38 | 74 | 351
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 15 | 21 | 25 | 23 | 16 | 23 | 124
  >=65 years | 1 | 30 | 24 | 48 | 51 | 22 | 51 | 227
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 2 | 45 | 45 | 73 | 74 | 38 | 74 | 351
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 3
  Not Hispanic or Latino | 2 | 40 | 40 | 53 | 56 | 28 | 51 | 270
  Unknown or Not Reported | 0 | 5 | 5 | 19 | 18 | 9 | 22 | 78
Race/Ethnicity, Customized [Number; unit: Participants] — Race
  Participants
    White | 2 | 33 | 37 | 70 | 72 | 32 | 67 | 313
    Black or African American | 0 | 6 | 3 | 2 | 2 | 5 | 6 | 24
    Other | 0 | 5 | 5 | 1 | 0 | 1 | 1 | 13
    Asian | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) Cohorts B and C Per BICR
Description: Objective response rate (ORR) is defined as the percent of participants who had confirmed complete or partial best overall response (BOR) per retrospective Blinded Independent Central Review (BICR) among treated participants with measurable disease at baseline. For participants without documented progression by RECIST v1.1 or subsequent therapy, all available response assessments contributed to the BOR assessment.
  Partial Response is at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Complete Response is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  Tumor assessments were performed every 8 weeks (± 7 days) for 6 months since treatment initiation and thereafter every 12 weeks (± 7 days).
  Confidence-interval based on Clopper Pearson method.
Time Frame: From first dose to the date of objectively documented progression or the date of subsequent systemic anti-cancer therapy, whichever occurred first (assessed up to approximately 61 months)
Population: All treated Cohort B and C participants with measurable disease at baseline; pre-specified only to be collected for Cohorts B and C.
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Cohort B: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg | Cohort C: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg
Number analyzed (Participants) | 32 | 30
Percent of Participants | 12.5 [3.5 to 29.0] | 20.0 [7.7 to 38.6]

2. Primary Outcome: Objective Response Rate (ORR) Cohort D
Description: In Cohort D, ORR is defined as the percentage of participants who had confirmed complete or partial BOR by BICR among randomized subjects with measurable disease at baseline as entered in Interactive Response Technologies web-based system (IWRS). For participants without documented progression or subsequent therapy, all available response assessments will contribute to the BOR assessment.
  Partial Response is at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Complete Response is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  Tumor assessments were performed every 8 weeks (± 7 days) for 6 months since treatment initiation and thereafter every 12 weeks (± 7 days).
  Confidence-interval based on Clopper Pearson method.
Time Frame: From randomization to the date of objectively documented progression or the date of subsequent systemic anti-cancer therapy, whichever occurred first (assessed up to approximately 61 months)
Population: All randomized Cohort D participants with measurable disease at baseline. For Arm D3 and D4 crossover participants, the data prior to the first dose date received in Arm D1 is being reported in their originally assigned Arm.
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Cohort D Arm 1: Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg Q3W | Cohort D Arm 2: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg Q6W | Cohort D Arm 3: Ipilimumab 3 mg/kg | Cohort D Arm 4: Cabazitaxel 20 mg/m2 or 25 mg/m2 + Prednisone 10 mg
Number analyzed (Participants) | 45 | 46 | 23 | 45
Percent of Participants | 8.9 [2.5 to 21.2] | 15.2 [6.3 to 28.9] | 4.3 [0.1 to 21.9] | 11.1 [3.7 to 24.1]

3. Primary Outcome: Radiographic Progression Free Survival (rPFS) for Cohorts B and C Per BICR
Description: Radiographic progression-free survival (rPFS) is defined as the time between the date of first treatment and the first date of documented radiographic progression or death due to any cause, whichever occurs first.
  The following progressive diseases were collected, documented and assessed as below:
  Radiographic progression per retrospective Blinded Independent Central Review (BICR) assessment
  1. Bone disease progression by Prostate Cancer Working Group (PCWG2)
  2. Non-bone soft tissue disease progression by RECIST v1.1 Progressive disease is at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm (the appearance of one or more new lesions is also considered progression).
  Based on Kaplan-Meier estimates.
Time Frame: From first dose to the date of objectively documented progression or death due to any cause, whichever occurred first (assessed up to approximately 61 months)
Population: All treated Cohort B and C participants. (i) Participants who did not progress or die were censored on the date of their last evaluable tumor assessment (ie, bone scan, CT, MRI). (ii) Participants who did not have any on study tumor assessments and did not die were censored on their date of first treatment. Pre-specified only to be collected for Cohorts B and C.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort B: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg | Cohort C: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg
Number analyzed (Participants) | 45 | 45
Months | 7.59 [3.65 to 10.22] | 5.36 [2.92 to 7.66]

4. Primary Outcome: Radiographic Progression-Free Survival (rPFS) for Cohort D
Description: Radiographic progression-free survival (rPFS) is defined as the time between the date of randomization and the first date of documented progression per BICR or death due to any cause, whichever occurs first.
  The following progressive diseases were collected, documented and assessed as below:
  Radiographic progression per BICR assessment
  1. Bone disease progression by (Prostate Cancer Working Group) PCWG2
  2. Non-bone soft tissue disease progression by RECIST v1.1 Progressive disease is at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm (the appearance of one or more new lesions is also considered progression).
  Based on Kaplan-Meier estimates.
Time Frame: From randomization and the first date of documented progression or death due to any cause, whichever occurs first (assessed up to approximately 61 months)
Population: All randomized Cohort D participants (i) Participants who did not progress or die were censored on the date of their last evaluable tumor assessment (ie, bone scan, CT, MRI). (ii) Participants who did not have any on study tumor assessments and did not die were censored on their date of randomization. For Arm D3 and D4 crossover participants, the data prior to the first dose date received in Arm D1 is being reported in their originally assigned Arm.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort D Arm 1: Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg Q3W | Cohort D Arm 2: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg Q6W | Cohort D Arm 3: Ipilimumab 3 mg/kg | Cohort D Arm 4: Cabazitaxel 20 mg/m2 or 25 mg/m2 + Prednisone 10 mg
Number analyzed (Participants) | 73 | 74 | 38 | 74
Months | 3.94 [2.17 to 7.62] | 4.17 [3.32 to 5.59] | 3.48 [2.14 to 5.78] | 7.92 [5.55 to 9.33]

5. Secondary Outcome: Radiographic/Clinical Progression Free Survival (rcPFS) for Cohorts B and C
Description: Radiographic/clinical progression-free survival (rcPFS) is the time between first dose and first documented progression or death due to any cause, whichever occurred first.
  Radiographic progression per Investigator assessment:
  1. Bone disease progression by Prostate Cancer Working Group (PCWG2)
  2. Non-bone soft tissue disease progression by RECIST v1.1
  Clinical progression per investigator assessment:
  1. Need for palliative radiation therapy involving more than one site, OR
  2. Surgery of kyphoplasty to any neoplastic lesion, OR
  3. Cancer-associated clinical deterioration determined by treating physician. Progressive disease is at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm (the appearance of one or more new lesions is also considered progression).
  Based on Kaplan-Meier estimates.
Time Frame: as for outcome 3
Population: All treated Cohort B, C participants. (i) Participants who did not progress or die were censored on the date of their last evaluable tumor assessment (ie, bone scan, CT, MRI). (ii) Participants who did not have any on study tumor assessments and did not die were censored on their date of first treatment. Pre-specified only to be collected for Cohorts B and C.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort B: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg | Cohort C: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg
Number analyzed (Participants) | 45 | 45
Months | 4.34 [2.79 to 5.49] | 3.71 [2.10 to 4.04]

6. Secondary Outcome: Radiographic/Clinical Progression Free Survival (rcPFS) for Cohort D
Description: as for outcome 5
Time Frame: From randomization and the first date of documented progression or death due to any cause, whichever occurs first (assessed up to approximately 93 months)
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort D Arm 1: Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg Q3W | Cohort D Arm 2: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg Q6W | Cohort D Arm 3: Ipilimumab 3 mg/kg | Cohort D Arm 4: Cabazitaxel 20 mg/m2 or 25 mg/m2 + Prednisone 10 mg
Number analyzed (Participants) | 73 | 74 | 38 | 74
Months | 2.53 [2.10 to 3.22] | 3.78 [2.23 to 4.63] | 2.66 [2.04 to 3.71] | 5.85 [3.84 to 7.52]

7. Secondary Outcome: Overall Survival (OS) Cohorts B and C
Description: Overall survival (OS) is defined as the time from first treatment to the date of death from any cause. For participants who were alive, their survival time was censored at the last known alive date. Overall survival was censored for participants at the date of first treatment if they had no follow-up.
  Based on Kaplan-Meier estimates.
Time Frame: From first dose to the date of death due to any cause (assessed up to approximately 61 months)
Population: All treated participants in Cohorts B and C; pre-specified only to be collected for Cohorts B and C.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort B: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg | Cohort C: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg
Number analyzed (Participants) | 45 | 45
Months | 19.75 [13.90 to 23.56] | 15.21 [8.44 to 17.77]

8. Secondary Outcome: Overall Survival (OS) Cohort D
Description: Overall survival (OS) is defined as the time from randomization to the date of death from any cause. For participants who were alive, their survival time was censored at the last known alive date. Overall survival was censored for participants at the date of first treatment if they had no follow-up.
  Based on Kaplan-Meier estimates.
Time Frame: From randomization to the date of death due to any cause (assessed up to approximately 93 months)
Population: All randomized participants in Cohort D.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort D Arm 1: Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg Q3W | Cohort D Arm 2: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg Q6W | Cohort D Arm 3: Ipilimumab 3 mg/kg | Cohort D Arm 4: Cabazitaxel 20 mg/m2 or 25 mg/m2 + Prednisone 10 mg
Number analyzed (Participants) | 73 | 74 | 38 | 74
Months | 15.9 [13.14 to 19.29] | 14.46 [10.64 to 17.51] | 18.46 [10.28 to 25.69] | 15.15 [11.56 to 18.56]

9. Secondary Outcome: Prostate-Specific Antigen Response Rate (PSA-RR) Cohorts B and C
Description: The percent of participants with a 50% or greater decrease in prostate-specific antigen (PSA) from baseline to the lowest post-baseline PSA result. BBaseline evaluations or events are defined as evaluations or events that occur before the date and time of the first dose of study treatment. Evaluations on the same date and time of the first dose of study treatment were considered as baseline evaluations.
  Confidence-interval based on Clopper Pearson method.
Time Frame: From baseline to the date of objectively documented progression or death due to any cause, whichever occurred first (assessed up to approximately 61 months)
Population: All treated participants with PSA values at baseline and at least one postbaseline assessment in Cohorts B and C. Pre-specified only to be collected for Cohorts B and C.
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Cohort B: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg | Cohort C: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg
Number analyzed (Participants) | 34 | 40
Percent of Participants | 17.6 [6.8 to 34.5] | 10.0 [2.8 to 23.7]

10. Secondary Outcome: Prostate-Specific Antigen Response Rate (PSA-RR) Cohort D
Description: The percent of participants with a 50% or greater decrease in prostate-specific antigen (PSA) from baseline to the lowest post-baseline PSA result. Baseline evaluations or events are defined as evaluations or events that occur before the date and time of the first dose of study treatment. Evaluations on the same date and time of the first dose of study treatment were considered as baseline evaluations.
  Confidence-interval based on Clopper Pearson method.
Time Frame: From baseline to the date of objectively documented progression or death due to any cause, whichever occurred first (assessed up to approximately 93 months)
Population: All randomized participants with PSA values at baseline and at least one post-baseline assessment in Cohort D. For Arm D3 and D4 crossover participants, the data prior to the first dose date received in Arm D1 is being reported.
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Groups:
- Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg Q4W After Crossover From Arm D3: Arm D3 participants who progressed on or after treatment were eligible to crossover to Arm D1. Nivolumab 3 mg/kg in combination with ipilimumab 1 mg/kg every 3 weeks for up to 4 doses (Cycles 1 to 4), followed by nivolumab 480 mg administered every 4 weeks (Cycle 5 and beyond). Participants receiving maintenance nivolumab with ongoing disease control or with radiographic progression were permitted re-induction with the combination of ipilimumab and nivolumab at their original combination dose upon PSA progression or radiographic progression (whichever occured first). Treatment continued until disease progression, unacceptable toxicity, withdrawal of consent, 2-year maximum treatment duration, or the study ends, whichever occurred first.
- Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg Q4W After Crossover From Arm D4: Arm D4 participants who progressed on or after treatment were eligible to crossover to Arm D1. Nivolumab 3 mg/kg in combination with ipilimumab 1 mg/kg every 3 weeks for up to 4 doses (Cycles 1 to 4), followed by nivolumab 480 mg administered every 4 weeks (Cycle 5 and beyond). Participants receiving maintenance nivolumab with ongoing disease control or with radiographic progression were permitted re-induction with the combination of ipilimumab and nivolumab at their original combination dose upon PSA progression or radiographic progression (whichever occured first). Treatment continued until disease progression, unacceptable toxicity, withdrawal of consent, 2-year maximum treatment duration, or the study ends, whichever occurred first.
Arm/Group | Cohort D Arm 1: Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg Q3W | Cohort D Arm 2: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg Q6W | Cohort D Arm 3: Ipilimumab 3 mg/kg | Cohort D Arm 4: Cabazitaxel 20 mg/m2 or 25 mg/m2 + Prednisone 10 mg | Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg Q4W After Crossover From Arm D3 | Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg Q4W After Crossover From Arm D4
Number analyzed (Participants) | 66 | 66 | 37 | 71 | 13 | 23
Percent of Participants | 13.6 [6.4 to 24.3] | 18.2 [9.8 to 29.6] | 5.4 [0.7 to 18.2] | 23.9 [14.6 to 35.5] | 30.8 [9.1 to 61.4] | 17.4 [5.0 to 38.8]

11. Secondary Outcome: The Number of Participants Experiencing Adverse Events (AEs) in Cohorts A, B and C
Description: An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation in a participant administered study treatment and that does not necessarily have a causal relationship with this treatment.
Time Frame: From first dose to 30 days after last dose of study therapy (an average of 2.8 months assessed up to approximately 18.2 months)
Population: All treated participants in Cohorts A, B and C
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg | Cohort B: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg | Cohort C: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg
Number analyzed (Participants) | 2 | 45 | 45
Participants | 2 | 45 | 45

12. Secondary Outcome: The Number of Participants Experiencing Adverse Events (AEs) in Cohort D
Description: as for outcome 11
Time Frame: From first dose to 30 days after last dose of study therapy (an average of 6.19 months assessed up to approximately 26.8 months)
Population: All treated participants in Cohort D. For Arm D3 and D4 crossover participants, the data prior to the first dose date received in Arm D1 is being reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort D Arm 1: Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg Q3W | Cohort D Arm 2: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg Q6W | Cohort D Arm 3: Ipilimumab 3 mg/kg | Cohort D Arm 4: Cabazitaxel 20 mg/m2 or 25 mg/m2 + Prednisone 10 mg | Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg Q4W After Crossover From Arm D3 | Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg Q4W After Crossover From Arm D4
Number analyzed (Participants) | 73 | 73 | 38 | 72 | 13 | 27
Participants | 69 | 71 | 37 | 69 | 11 | 27

13. Secondary Outcome: The Number of Participants Experiencing Serious Adverse Events (SAEs) in Cohorts A, B and C
Description: A Serious Adverse Event (SAE) is defined as any untoward medical occurrence that at any dose results in death, is life-threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is an important medical event.
Time Frame: as for outcome 11
Population: All treated participants in Cohorts A, B and C
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg | Cohort B: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg | Cohort C: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg
Number analyzed (Participants) | 2 | 45 | 45
Participants | 1 | 17 | 33

14. Secondary Outcome: The Number of Participants Experiencing Serious Adverse Events (SAEs) in Cohort D
Description: as for outcome 13
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort D Arm 1: Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg Q3W | Cohort D Arm 2: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg Q6W | Cohort D Arm 3: Ipilimumab 3 mg/kg | Cohort D Arm 4: Cabazitaxel 20 mg/m2 or 25 mg/m2 + Prednisone 10 mg | Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg Q4W After Crossover From Arm D3 | Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg Q4W After Crossover From Arm D4
Number analyzed (Participants) | 73 | 73 | 38 | 72 | 13 | 27
Participants | 38 | 44 | 15 | 32 | 7 | 18

15. Secondary Outcome: The Number of Participants Experiencing Adverse Events (AEs) Leading to Discontinuation in Cohorts A, B and C
Description: An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered study treatment and that does not necessarily have a causal relationship with this treatment.
Time Frame: as for outcome 11
Population: All treated participants in Cohorts A, B and C
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg | Cohort B: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg | Cohort C: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg
Number analyzed (Participants) | 2 | 45 | 45
Participants | 1 | 17 | 18

16. Secondary Outcome: The Number of Participants Experiencing Adverse Events (AEs) Leading to Discontinuation in Cohort D
Description: as for outcome 15
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort D Arm 1: Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg Q3W | Cohort D Arm 2: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg Q6W | Cohort D Arm 3: Ipilimumab 3 mg/kg | Cohort D Arm 4: Cabazitaxel 20 mg/m2 or 25 mg/m2 + Prednisone 10 mg | Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg Q4W After Crossover From Arm D3 | Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg Q4W After Crossover From Arm D4
Number analyzed (Participants) | 73 | 73 | 38 | 72 | 13 | 27
Participants | 16 | 27 | 7 | 13 | 3 | 6

17. Secondary Outcome: The Number of Participants Experiencing Immune Mediated Adverse Events in Cohorts A, B and C
Description: Immune-mediated adverse events (IMAEs) are AEs consistent with an immune-mediated mechanism or immune-mediated component for which non-inflammatory etiologies (eg, infection or tumor progression) have been ruled out. IMAEs can include events with an alternate etiology which were exacerbated by the induction of autoimmunity.
Time Frame: From first dose to 100 days after last dose of study therapy (an average of 2.8 months assessed up to approximately 20.7 months)
Population: All treated participants in Cohorts A, B and C.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg | Cohort B: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg | Cohort C: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg
Number analyzed (Participants) | 2 | 45 | 45
Participants
  Pneumonitis | 1 | 3 | 2
  Diarrhea/Colitis | 0 | 15 | 17
  Hepatitis | 0 | 4 | 1
  Adrenal Insufficiency | 0 | 1 | 2
  Hypothyroidism/Thyroiditis | 0 | 2 | 1
  Diabetes Mellitus | 0 | 0 | 0
  Nephritis and Renal Dysfunction | 0 | 1 | 0
  Rash | 0 | 16 | 6
  Hypersensitivity | 0 | 0 | 0
  Hyperthyroidism | 0 | 1 | 1
  Hypophysitis | 0 | 3 | 1

18. Secondary Outcome: The Number of Participants Experiencing Immune Mediated Adverse Events in Cohort D
Description: as for outcome 17
Time Frame: From first dose to 100 days after last dose of study therapy (an average of 8.48 months assessed up to approximately 29.09 months)
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort D Arm 1: Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg Q3W | Cohort D Arm 2: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg Q6W | Cohort D Arm 3: Ipilimumab 3 mg/kg | Cohort D Arm 4: Cabazitaxel 20 mg/m2 or 25 mg/m2 + Prednisone 10 mg | Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg Q4W After Crossover From Arm D3 | Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg Q4W After Crossover From Arm D4
Number analyzed (Participants) | 73 | 73 | 38 | 72 | 13 | 27
Participants
  Pneumonitis | 1 | 4 | 0 | 0 | 1 | 2
  Diarrhea/Colitis | 9 | 21 | 5 | 0 | 0 | 2
  Hepatitis | 5 | 8 | 0 | 0 | 0 | 2
  Adrenal Insufficiency | 2 | 3 | 1 | 0 | 2 | 1
  Hypothyroidism/Thyroiditis | 6 | 9 | 1 | 0 | 3 | 3
  Diabetes Mellitus | 1 | 1 | 0 | 0 | 0 | 1
  Nephritis and Renal Dysfunction | 0 | 0 | 0 | 0 | 0 | 0
  Rash | 12 | 10 | 2 | 0 | 1 | 4
  Hypersensitivity | 0 | 0 | 0 | 0 | 0 | 0
  Hyperthyroidism | 4 | 5 | 0 | 0 | 1 | 2
  Hypophysitis | 2 | 5 | 3 | 0 | 1 | 1

19. Secondary Outcome: The Number of Participants Who Died in Cohorts A, B and C
Description: Death due to any cause.
Time Frame: as for outcome 17
Population: All treated participants in Cohorts A, B and C.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg | Cohort B: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg | Cohort C: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg
Number analyzed (Participants) | 2 | 45 | 45
Participants | 2 | 39 | 39

20. Secondary Outcome: The Number of Participants Who Died in Cohort D
Description: Death due to any cause.
Time Frame: as for outcome 18
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort D Arm 1: Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg Q3W | Cohort D Arm 2: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg Q6W | Cohort D Arm 3: Ipilimumab 3 mg/kg | Cohort D Arm 4: Cabazitaxel 20 mg/m2 or 25 mg/m2 + Prednisone 10 mg | Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg Q4W After Crossover From Arm D3 | Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg Q4W After Crossover From Arm D4
Number analyzed (Participants) | 73 | 73 | 38 | 72 | 13 | 27
Participants | 14 | 15 | 4 | 13 | 2 | 9

21. Secondary Outcome: The Number of Participants With Changes in Laboratory Values From Baseline in Cohorts A, B and C
Description: The number of participants with a change in laboratory values from baseline Grade in Cohorts A, B and C.
Time Frame: as for outcome 11
Population: All treated participants in Cohorts A, B and C with baseline laboratory measurements.
Measure: Number; unit: Participants
Arm/Group | Cohort A: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg | Cohort B: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg | Cohort C: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg
Number analyzed (Participants) | 2 | 33 | 45
Participants
  Hemoglobin: number analyzed (Participants) | 1 | 31 | 43
  Hemoglobin | 0 | 6 | 23
  Platelet Count: number analyzed (Participants) | 1 | 30 | 43
  Platelet Count | 0 | 3 | 8
  Leukocytes: number analyzed (Participants) | 1 | 30 | 44
  Leukocytes | 0 | 1 | 7
  Lymphocytes (Absolute): number analyzed (Participants) | 1 | 30 | 43
  Lymphocytes (Absolute) | 0 | 9 | 17
  Absolute Neutrophil Count: number analyzed (Participants) | 1 | 30 | 43
  Absolute Neutrophil Count | 0 | 0 | 6
  Alkaline Phosphatase: number analyzed (Participants) | 1 | 29 | 40
  Alkaline Phosphatase | 0 | 7 | 15
  Aspartate Aminotransferase: number analyzed (Participants) | 1 | 29 | 43
  Aspartate Aminotransferase | 0 | 9 | 17
  Alanine Aminotransferase: number analyzed (Participants) | 1 | 30 | 43
  Alanine Aminotransferase | 1 | 5 | 14
  Bilirubin, Total: number analyzed (Participants) | 1 | 30 | 43
  Bilirubin, Total | 0 | 3 | 0
  Creatinine: number analyzed (Participants) | 1 | 30 | 43
  Creatinine | 0 | 5 | 8
  Amylase, Total: number analyzed (Participants) | 1 | 30 | 41
  Amylase, Total | 0 | 8 | 6
  Lipase, Total: number analyzed (Participants) | 1 | 30 | 40
  Lipase, Total | 0 | 6 | 3
  Hypernatremia: number analyzed (Participants) | 1 | 30 | 41
  Hypernatremia | 0 | 1 | 0
  Hyponatremia: number analyzed (Participants) | 1 | 30 | 41
  Hyponatremia | 0 | 8 | 15
  Hyperkalemia: number analyzed (Participants) | 1 | 30 | 42
  Hyperkalemia | 0 | 1 | 5
  Hypokalemia: number analyzed (Participants) | 1 | 30 | 42
  Hypokalemia | 0 | 3 | 7
  Hypercalcemia: number analyzed (Participants) | 1 | 29 | 41
  Hypercalcemia | 0 | 0 | 0
  Hypocalcemia: number analyzed (Participants) | 1 | 29 | 41
  Hypocalcemia | 0 | 4 | 12
  Hyperglycemia: number analyzed (Participants) | 0 | 2 | 4
  Hyperglycemia |  | 0 | 2
  Hypoglycemia: number analyzed (Participants) | 0 | 2 | 42
  Hypoglycemia |  | 0 | 0

22. Secondary Outcome: The Number of Participants With Changes in Laboratory Values From Baseline in Cohort D
Description: The number of participants with an change in laboratory values from baseline Grade in Cohort D.
Time Frame: as for outcome 12
Population: All treated participants in Cohort D with baseline laboratory measurements. For Arm D3 and D4 crossover participants, the data prior to the first dose date received in Arm D1 is being reported in their originally assigned Arm.
Measure: Number; unit: Participants
Arm/Group | Cohort D Arm 1: Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg Q3W | Cohort D Arm 2: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg Q6W | Cohort D Arm 3: Ipilimumab 3 mg/kg | Cohort D Arm 4: Cabazitaxel 20 mg/m2 or 25 mg/m2 + Prednisone 10 mg
Number analyzed (Participants) | 71 | 67 | 37 | 71
Participants
  Hemoglobin: number analyzed (Participants) | 70 | 66 | 37 | 71
  Hemoglobin | 26 | 35 | 14 | 42
  Platelet Count: number analyzed (Participants) | 70 | 65 | 37 | 71
  Platelet Count | 10 | 8 | 2 | 15
  Leukocytes: number analyzed (Participants) | 70 | 66 | 37 | 71
  Leukocytes | 8 | 9 | 3 | 25
  Lymphocytes (Absolute): number analyzed (Participants) | 70 | 64 | 37 | 71
  Lymphocytes (Absolute) | 28 | 31 | 9 | 37
  Absolute Neutrophil Count: number analyzed (Participants) | 70 | 65 | 37 | 71
  Absolute Neutrophil Count | 7 | 7 | 2 | 18
  Alkaline Phosphatase: number analyzed (Participants) | 71 | 65 | 37 | 71
  Alkaline Phosphatase | 23 | 18 | 12 | 14
  Aspartate Aminotransferase: number analyzed (Participants) | 68 | 65 | 37 | 71
  Aspartate Aminotransferase | 17 | 21 | 5 | 11
  Alanine Aminotransferase: number analyzed (Participants) | 71 | 65 | 37 | 71
  Alanine Aminotransferase | 21 | 24 | 3 | 6
  Bilirubin, Total: number analyzed (Participants) | 71 | 65 | 37 | 71
  Bilirubin, Total | 3 | 1 | 0 | 3
  Creatinine | 20 | 15 | 2 | 14
  Amylase, Total: number analyzed (Participants) | 55 | 56 | 32 | 63
  Amylase, Total | 13 | 16 | 1 | 3
  Lipase, Total: number analyzed (Participants) | 67 | 60 | 37 | 69
  Lipase, Total | 17 | 16 | 7 | 8
  Hypernatremia: number analyzed (Participants) | 71 | 66 | 37 | 71
  Hypernatremia | 4 | 4 | 1 | 3
  Hyponatremia: number analyzed (Participants) | 71 | 66 | 37 | 71
  Hyponatremia | 21 | 12 | 7 | 12
  Hyperkalemia: number analyzed (Participants) | 70 | 66 | 37 | 70
  Hyperkalemia | 7 | 12 | 1 | 7
  Hypokalemia: number analyzed (Participants) | 70 | 66 | 37 | 70
  Hypokalemia | 5 | 8 | 5 | 8
  Hypercalcemia: number analyzed (Participants) | 68 | 64 | 37 | 69
  Hypercalcemia | 2 | 7 | 2 | 1
  Hypocalcemia: number analyzed (Participants) | 68 | 64 | 37 | 69
  Hypocalcemia | 12 | 23 | 14 | 18
  Hyperglycemia: number analyzed (Participants) | 13 | 17 | 6 | 17
  Hyperglycemia | 1 | 9 | 3 | 5
  Hypoglycemia: number analyzed (Participants) | 13 | 17 | 6 | 17
  Hypoglycemia | 0 | 0 | 0 | 1

23. Secondary Outcome: The Number of Participants With Liver Function Laboratory Abnormalities in Cohorts A, B and C
Description: The number of participants with laboratory abnormalities in specific liver tests based on SI conventional units.
  ALT = Alanine Aminotransferase AST = Aspartate Aminotransferase ULN = Upper Limit of Normal
Time Frame: as for outcome 11
Population: All Treated Participants in Cohorts A, B and C with at least one on-treatment liver function measurement.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg | Cohort B: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg | Cohort C: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg
Number analyzed (Participants) | 1 | 31 | 43
Participants
  ALT OR AST > 3XULN | 0 | 2 | 5
  ALT OR AST> 5XULN | 0 | 2 | 2
  ALT OR AST> 10XULN | 0 | 2 | 1
  ALT OR AST > 20XULN | 0 | 2 | 1
  TOTAL BILIRUBIN > 2XULN | 0 | 2 | 0

24. Secondary Outcome: The Number of Participants With Liver Function Laboratory Abnormalities in Cohort D
Description: as for outcome 23
Time Frame: as for outcome 12
Population: All Treated Participants in Cohort D with at least one on-treatment liver function measurement. For Arm D3 and D4 crossover participants, the data prior to the first dose date received in Arm D1 is being reported in their originally assigned Arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort D Arm 1: Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg Q3W | Cohort D Arm 2: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg Q6W | Cohort D Arm 3: Ipilimumab 3 mg/kg | Cohort D Arm 4: Cabazitaxel 20 mg/m2 or 25 mg/m2 + Prednisone 10 mg
Number analyzed (Participants) | 71 | 65 | 37 | 71
Participants
  ALT OR AST > 3XULN | 6 | 8 | 0 | 1
  ALT OR AST> 5XULN | 3 | 5 | 0 | 0
  ALT OR AST> 10XULN | 1 | 3 | 0 | 0
  ALT OR AST > 20XULN | 0 | 1 | 0 | 0
  TOTAL BILIRUBIN > 2XULN | 2 | 0 | 0 | 0
  ALP>1.5XULN | 23 | 24 | 15 | 17
  CONCURR ALT/ AST ELEV>3XULN WITH TOT BILI>1.5XULN WITHIN 1 DAY | 1 | 0 | 0 | 0
  CONCURR ALT/ AST ELEV>3XULN WITH TOT BILI>1.5XULN WITHIN 30 DAYS | 1 | 0 | 0 | 0
  CONCURR ALT/ AST ELEV>3XULN WITH TOT BILI>2XULN WITHIN 1 DAY | 1 | 0 | 0 | 0
  CONCURR ALT/ AST ELEV>3XULN WITH TOT BILI>2XULN WITHIN 30 DAYS | 1 | 0 | 0 | 0

25. Secondary Outcome: The Number of Participants With Thyroid Function Laboratory Abnormalities in Cohort A, B and C
Description: The number of participants with laboratory abnormalities in specific thyroid tests based on SI conventional units.
  TSH = Thyroid Stimulating Hormone LLN = Lower Limit of Normal ULN = Upper Limit of Normal
Time Frame: as for outcome 11
Population: Treated participants in Cohorts A, B and C with at least one on-treatment TSH measurement. Treated subjects in Cohort B with adequate follow-up of at least 24 weeks are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg | Cohort B: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg | Cohort C: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg
Number analyzed (Participants) | 1 | 29 | 41
Participants
  TSH > ULN | 0 | 5 | 13
  TSH > ULN WITH TSH <= ULN AT BASELINE | 0 | 3 | 7
  TSH >ULN WITH ATLEAST ONE FT3/FT4 TEST VALUE <LLN | 0 | 4 | 6
  TSH >ULN WITH ALL OTHER FT3/FT4 TEST VALUES >= LLN | 0 | 1 | 4
  TSH > ULN WITH FT3/FT4 TEST MISSING | 0 | 0 | 3
  TSH < LLN | 0 | 7 | 10
  TSH <LLN WITH TSH >= LLN AT BASELINE | 0 | 6 | 10
  TSH <LLN WITH ATLEAST ONE FT3/FT4 TEST VALUE > ULN | 0 | 4 | 8
  TSH <LLN WITH ALL OTHER FT3/FT4 TEST VALUES <= ULN | 0 | 2 | 1
  TSH < LLN WITH FT3/FT4 TEST MISSING | 0 | 1 | 1

26. Secondary Outcome: The Number of Participants With Thyroid Function Laboratory Abnormalities in Cohort D
Description: as for outcome 25
Time Frame: as for outcome 12
Population: Treated participants in Cohort D with at least one on-treatment TSH measurement. For Arm D3 and D4 crossover participants, the data prior to the first dose date received in Arm D1 is being reported in their originally assigned Arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort D Arm 1: Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg Q3W | Cohort D Arm 2: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg Q6W | Cohort D Arm 3: Ipilimumab 3 mg/kg | Cohort D Arm 4: Cabazitaxel 20 mg/m2 or 25 mg/m2 + Prednisone 10 mg
Number analyzed (Participants) | 70 | 62 | 37 | 71
Participants
  TSH > ULN | 13 | 20 | 1 | 11
  TSH > ULN WITH TSH <= ULN AT BASELINE | 10 | 16 | 1 | 6
  TSH >ULN WITH ATLEAST ONE FT3/FT4 TEST VALUE <LLN | 6 | 12 | 0 | 3
  TSH >ULN WITH ALL OTHER FT3/FT4 TEST VALUES >= LLN | 6 | 7 | 1 | 5
  TSH > ULN WITH FT3/FT4 TEST MISSING | 1 | 1 | 0 | 3
  TSH < LLN | 22 | 22 | 7 | 6
  TSH <LLN WITH TSH >= LLN AT BASELINE | 22 | 20 | 6 | 5
  TSH <LLN WITH ATLEAST ONE FT3/FT4 TEST VALUE > ULN | 9 | 9 | 1 | 3
  TSH <LLN WITH ALL OTHER FT3/FT4 TEST VALUES <= ULN | 13 | 11 | 5 | 3
  TSH < LLN WITH FT3/FT4 TEST MISSING | 0 | 2 | 1 | 0

27. Secondary Outcome: Changes in Pain Severity as Measured by the Brief Pain Inventory-Short Form (BPI-SF) Scores Cohorts B and C
Description: Change between Mean BPI-SF scores at baseline and week 4 (cycle 2). The BPI-SF measures pain severity through the use of a numerical rating scale. Participants rate the severity of their pain at its ''worst,'' ''least,'' and ''average'' in the last 24 hours using an 11-point numerical rating scale with anchors of ''0 = no pain'' and ''10 = pain as bad as you can imagine.'' A higher score = a "worse" outcome. Pain Severity Score = Mean of items 3-6 (pain at its worst, pain at its least). Baseline evaluations or events are defined as evaluations or events that occur before the date and time of the first dose of study treatment. Evaluations on the same date and time of the first dose of study treatment were considered as baseline evaluations.
Time Frame: At baseline and Week 4 (Cycle 2)
Population: All treated Cohort B and C participants with baseline and week 4 (cycle 2) scores. Pre-specified only to be collected for Cohorts B and C.
Measure: Mean (Full Range); unit: Score on a scale
Arm/Group | Cohort B: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg | Cohort C: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg
Number analyzed (Participants) | 21 | 29
Score on a scale
  Worst pain in the last 24 hours Week 4 (Cycle 2) | 0.0 [-4 to 5] | -0.1 [-5 to 6]
  Least pain in the last 24 hours Week 4 (Cycle 2): number analyzed (Participants) | 20 | 29
  Least pain in the last 24 hours Week 4 (Cycle 2) | -0.5 [-3 to 1] | -0.1 [-3 to 3]
  Average pain in the last 24 hours Week 4 (Cycle 2): number analyzed (Participants) | 19 | 29
  Average pain in the last 24 hours Week 4 (Cycle 2) | -0.2 [-3 to 2] | -0.1 [-4 to 2]
  Current pain Week 4 (Cycle 2): number analyzed (Participants) | 20 | 29
  Current pain Week 4 (Cycle 2) | -0.1 [-3 to 2] | 0 [-5 to 4]

28. Secondary Outcome: Changes in Pain Severity as Measured by the Brief Pain Inventory-Short Form (BPI-SF) Scores Cohort D
Description: as for outcome 27
Time Frame: At baseline and 4 weeks after first dose.
Population: All randomized Cohort D participants with baseline and week 4 scores
Measure: Mean (Full Range); unit: Score on a scale
Arm/Group | Cohort D Arm 1: Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg Q3W | Cohort D Arm 2: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg Q6W | Cohort D Arm 3: Ipilimumab 3 mg/kg | Cohort D Arm 4: Cabazitaxel 20 mg/m2 or 25 mg/m2 + Prednisone 10 mg
Number analyzed (Participants) | 54 | 47 | 34 | 61
Score on a scale
  Worst pain in the last 24 hours Week 4: number analyzed (Participants) | 54 | 46 | 34 | 61
  Worst pain in the last 24 hours Week 4 | -0.3 [-7 to 8] | 0.5 [-5 to 7] | -0.1 [-8 to 6] | -0.5 [-7 to 5]
  Least pain in the last 24 hours Week 4: number analyzed (Participants) | 53 | 46 | 32 | 61
  Least pain in the last 24 hours Week 4 | -0.3 [-7 to 8] | 0.2 [-4 to 4] | 0.2 [-4 to 5] | -0.3 [-5 to 3]
  Average pain in the last 24 hours Week 4: number analyzed (Participants) | 52 | 46 | 32 | 61
  Average pain in the last 24 hours Week 4 | -0.5 [-6 to 6] | 0.2 [-5 to 6] | -0.3 [-5 to 5] | -0.4 [-5 to 3]
  Current pain Week 4: number analyzed (Participants) | 51 | 47 | 32 | 61
  Current pain Week 4 | -0.2 [-6 to 6] | 0.3 [-4 to 4] | -0.4 [-6 to 6] | -0.3 [-6 to 5]

29. Secondary Outcome: Change in Cancer-Related Symptoms and Quality of Life (QoL) by Functional Assessment of Cancer Therapy - Prostate (FACT-P) Questionnaire Cohort D
Description: The Functional Assessment of Cancer Therapy - Prostate (FACT-P) is a multidimensional, self-report Quality of Life (QoL) instrument designed for use with prostate cancer patients. It consists of 27 core items. The Functional Assessment of Cancer Therapy - General (FACT-G) questionnaire, which assesses patient function in 4 domains: Physical, Social/Family, Emotional, and Functional well-being. This is further supplemented by the Prostate Cancer Subscale (PCS), 12 disease-specific items to assess for prostate-related symptoms. Each item is rated from 0 (Not at all) to 4 (Very much) and combined to produce subscale scores for each domain, a Trial Outcome Index which is based on the Physical and Functional well-being scales and the PCS as well as a total score which ranges from 0 to 156. Higher scores represent better QoL. Baseline evaluations or events were defined as those that occur before or on the date and time of the first dose of study treatment.
Time Frame: At baseline and 4 weeks after first dose.
Population: All randomized Cohort D participants with baseline and week 4 scores; pre-specified for data to be collected only from Cohort D participants.
Measure: Mean (Full Range); unit: Score on a scale
Arm/Group | Cohort D Arm 1: Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg Q3W | Cohort D Arm 2: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg Q6W | Cohort D Arm 3: Ipilimumab 3 mg/kg | Cohort D Arm 4: Cabazitaxel 20 mg/m2 or 25 mg/m2 + Prednisone 10 mg
Number analyzed (Participants) | 57 | 48 | 35 | 64
Score on a scale | 6.73 [-60.2 to 116.4] | -4.74 [-81.0 to 72.7] | -3.64 [-91.5 to 65] | -0.28 [-71.7 to 53.0]

30. Secondary Outcome: Change From Baseline in Health Status and Health Utility by 3-level EuroQol Five Dimensions (EQ-5D-3L) Questionnaire Cohorts B and C
Description: The European Quality of Life 5D-3L Scale (EQ-5D-3L) assesses general health-related quality of life. Health is defined in 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems. Responses are: '1' = no problem, and '3' = the most serious problem. The responses are combined in a 5-digit number. These health states are converted to a single index value using the crosswalk method to the EQ-5D-3L value set from the United Kingdom (UK). The EQ-5D-3L health utility index based on the UK population weights range from -0.594 to 1.0 with higher scores indicating higher health utility. Baseline evaluations or events are defined as occurring before the date and time of the first dose of study treatment. Evaluations on the same date and time of the first dose of study treatment were considered as baseline evaluations.
Time Frame: At baseline and at Week 4 of Cycle 2.
Population: as for outcome 27
Measure: Mean (Full Range); unit: Score on a scale
Arm/Group | Cohort B: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg | Cohort C: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg
Number analyzed (Participants) | 20 | 26
Score on a scale | 0.0083 [-0.311 to 0.275] | -0.0074 [-0.327 to 0.628]

31. Secondary Outcome: Change From Baseline in Health Status and Health Utility by 3-level EuroQol Five Dimensions (EQ-5D-3L) Questionnaire Cohort D
Description: as for outcome 30
Time Frame: At baseline and 4 weeks after first dose.
Population: All randomized Cohort D participants with baseline and week 4 scores
Measure: Mean (Full Range); unit: Score on a scale
Arm/Group | Cohort D Arm 1: Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg Q3W | Cohort D Arm 2: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg Q6W | Cohort D Arm 3: Ipilimumab 3 mg/kg | Cohort D Arm 4: Cabazitaxel 20 mg/m2 or 25 mg/m2 + Prednisone 10 mg
Number analyzed (Participants) | 54 | 45 | 33 | 62
Score on a scale | 0.0032 [-0.736 to 0.791] | -0.0328 [-0.574 to 0.532] | 0.0113 [-0.532 to 0.463] | 0.0219 [-0.514 to 0.697]

32. Post Hoc Outcome: Objective Response Rate (ORR) Cohort D
Description: as for outcome 2
Time Frame: From randomization to the date of objectively documented progression or the date of subsequent systemic anti-cancer therapy, whichever occurred first (assessed up to approximately 93 months)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Cohort D Arm 1: Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg Q3W | Cohort D Arm 2: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg Q6W | Cohort D Arm 3: Ipilimumab 3 mg/kg | Cohort D Arm 4: Cabazitaxel 20 mg/m2 or 25 mg/m2 + Prednisone 10 mg
Number analyzed (Participants) | 45 | 46 | 23 | 45
Percent of Participants | 13.3 [5.1 to 26.8] | 17.4 [7.8 to 31.4] | 8.7 [1.1 to 28.0] | 8.9 [2.5 to 21.2]

33. Post Hoc Outcome: Radiographic Progression-Free Survival (rPFS) for Cohort D
Description: as for outcome 4
Time Frame: as for outcome 6
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort D Arm 1: Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg Q3W | Cohort D Arm 2: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg Q6W | Cohort D Arm 3: Ipilimumab 3 mg/kg | Cohort D Arm 4: Cabazitaxel 20 mg/m2 or 25 mg/m2 + Prednisone 10 mg
Number analyzed (Participants) | 73 | 74 | 38 | 74
Months | 3.70 [2.37 to 5.36] | 3.81 [2.23 to 4.63] | 3.09 [2.04 to 4.37] | 6.34 [5.22 to 8.31]

ADVERSE EVENTS:
Time Frame: Participants will be assessed for All-Cause Mortality (ACM) from the date of their first dose of study therapy until study completion for Cohorts A, B and C and from randomization until study completion for Cohort D (assessed up to approximately 93 months). SAEs and Other AEs were assessed from first dose to 100 days after last dose of study therapy for all Cohorts (assessed up to approximately 29.09 months).
Description: The number at Risk for ACM represents all Treated Participants in Cohorts A, B and C and all Randomized Participants in Cohort D. The at Risk for Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medicine for all Cohorts. For Arm D3 and D4 crossover, data prior to the first dose date received in Arm D1 is also being reported in their originally assigned Arm. Data are collected per cohort as prespecified.
Arm/Group | Cohort A: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg | Cohort B: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg | Cohort C: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg | Cohort D Arm 1: Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg Q3W | Cohort D Arm 2: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg Q6W | Cohort D Arm 3: Ipilimumab 3 mg/kg | Cohort D Arm 4: Cabazitaxel 20 mg/m2 or 25 mg/m2 + Prednisone 10 mg | Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg Q4W After Crossover From Arm D3 | Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg Q4W After Crossover From Arm D4
All-Cause Mortality (participants affected / at risk) | 2/2 | 40/45 | 41/45 | 67/73 | 65/74 | 28/38 | 49/74 | 9/13 | 21/27
Serious Adverse Events (participants affected / at risk) | 2/2 | 37/45 | 39/45 | 44/73 | 50/73 | 25/38 | 50/72 | 9/13 | 20/27
Other Adverse Events (participants affected / at risk) | 2/2 | 44/45 | 45/45 | 66/73 | 64/73 | 37/38 | 71/72 | 10/13 | 25/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg (N=2) | Cohort B: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg (N=45) | Cohort C: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg (N=45) | Cohort D Arm 1: Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg Q3W (N=73) | Cohort D Arm 2: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg Q6W (N=73) | Cohort D Arm 3: Ipilimumab 3 mg/kg (N=38) | Cohort D Arm 4: Cabazitaxel 20 mg/m2 or 25 mg/m2 + Prednisone 10 mg (N=72) | Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg Q4W After Crossover From Arm D3 (N=13) | Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg Q4W After Crossover From Arm D4 (N=27)
Agranulocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 3 | 0 | 3 | 3 | 2 | 6 | 1 | 2
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 3 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 4 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Myocarditis (Cardiac disorders) | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 2 | 1 | 0 | 0 | 2 | 0 | 2 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Hypophysitis (Endocrine disorders) | 0 | 0 | 1 | 1 | 2 | 3 | 0 | 1 | 0
Hypopituitarism (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Immune-mediated hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Thyroiditis (Endocrine disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Autoimmune colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 5 | 9 | 3 | 7 | 1 | 2 | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 7 | 5 | 6 | 2 | 4 | 0 | 2
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 6 | 2 | 0 | 0 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Large intestinal ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 1
Obstructive pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Overflow diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatolithiasis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 2
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Terminal ileitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 3 | 0 | 2 | 0 | 1 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 2 | 1 | 1 | 0 | 2 | 0 | 1
Death (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Fatigue (General disorders) | 0 | 2 | 3 | 0 | 2 | 0 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 2 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pain (General disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 1 | 4 | 2 | 2 | 2 | 0 | 1
Sudden death (General disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Brain abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cytomegalovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cytomegalovirus infection reactivation (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diarrhoea infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1
Eye infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Kidney infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenic infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 5 | 1 | 2 | 1 | 1 | 0
Rectal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 2 | 0 | 3 | 1 | 1 | 1
Septic shock (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Skin infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 3 | 3 | 1 | 1
Urosepsis (Infections and infestations) | 0 | 0 | 1 | 1 | 2 | 0 | 1 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Craniofacial fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Nerve root injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Shoulder fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood urine present (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Platelet count decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Troponin T increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 2 | 1 | 2 | 1 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 2 | 0 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 1 | 1 | 1 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Joint neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 3 | 11 | 8 | 3 | 18 | 2 | 6
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Brain oedema (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Cerebellar stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 2 | 2 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Embolic stroke (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Facial paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Guillain-Barre syndrome (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Immune-mediated encephalitis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Myasthenia gravis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraparesis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 1 | 1 | 2 | 2 | 3 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 4 | 3 | 2 | 3 | 0 | 0 | 0 | 0
Bladder neck obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bladder obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 4 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 3 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Ureteric stenosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Autoimmune lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diaphragmalgia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 1 | 0 | 1 | 2 | 1 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 3 | 1 | 4 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Circulatory collapse (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Iliac vein occlusion (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg (N=2) | Cohort B: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg (N=45) | Cohort C: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg (N=45) | Cohort D Arm 1: Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg Q3W (N=73) | Cohort D Arm 2: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg Q6W (N=73) | Cohort D Arm 3: Ipilimumab 3 mg/kg (N=38) | Cohort D Arm 4: Cabazitaxel 20 mg/m2 or 25 mg/m2 + Prednisone 10 mg (N=72) | Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg Q4W After Crossover From Arm D3 (N=13) | Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg Q4W After Crossover From Arm D4 (N=27)
Anaemia (Blood and lymphatic system disorders) | 1 | 13 | 14 | 10 | 15 | 9 | 26 | 4 | 6
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 8 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 3 | 1 | 5 | 1 | 1
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 2 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 3 | 0 | 4 | 0 | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 3 | 1 | 2 | 2 | 2 | 1 | 1
Addison's disease (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 1 | 1 | 2 | 2 | 2 | 1 | 1 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 2 | 4 | 4 | 5 | 1 | 2 | 0 | 2
Hypophysitis (Endocrine disorders) | 0 | 3 | 1 | 2 | 4 | 2 | 1 | 0 | 1
Hypothyroidism (Endocrine disorders) | 1 | 6 | 9 | 5 | 9 | 3 | 4 | 2 | 3
Dry eye (Eye disorders) | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 1 | 0
Eyelid haematoma (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Vision blurred (Eye disorders) | 1 | 2 | 5 | 1 | 2 | 1 | 3 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 4 | 4 | 3 | 0 | 2 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 7 | 4 | 6 | 4 | 4 | 3 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 2 | 0
Colitis (Gastrointestinal disorders) | 0 | 3 | 6 | 0 | 5 | 1 | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 17 | 15 | 13 | 7 | 11 | 20 | 1 | 4
Diarrhoea (Gastrointestinal disorders) | 0 | 23 | 28 | 24 | 26 | 15 | 24 | 4 | 5
Dry mouth (Gastrointestinal disorders) | 0 | 7 | 6 | 3 | 2 | 3 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 4 | 3 | 0 | 1 | 6 | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 3 | 0 | 5 | 0 | 1
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 6 | 2 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 13 | 19 | 18 | 17 | 9 | 28 | 2 | 8
Oral pain (Gastrointestinal disorders) | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 2 | 1 | 0 | 1 | 4 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 8 | 16 | 12 | 10 | 4 | 12 | 1 | 4
Asthenia (General disorders) | 0 | 4 | 7 | 6 | 5 | 6 | 11 | 1 | 5
Fatigue (General disorders) | 1 | 28 | 31 | 21 | 20 | 15 | 31 | 1 | 5
Gait disturbance (General disorders) | 0 | 0 | 3 | 2 | 0 | 1 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 3 | 1 | 1 | 4 | 1 | 1
Non-cardiac chest pain (General disorders) | 0 | 1 | 1 | 1 | 0 | 1 | 2 | 1 | 0
Oedema peripheral (General disorders) | 0 | 8 | 6 | 4 | 7 | 7 | 11 | 1 | 4
Pain (General disorders) | 0 | 5 | 3 | 9 | 4 | 1 | 10 | 0 | 4
Pyrexia (General disorders) | 1 | 9 | 14 | 7 | 6 | 6 | 8 | 1 | 4
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 3 | 2 | 2 | 1 | 2
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 0
Extradural abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Intervertebral discitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 2 | 1 | 4 | 2 | 1 | 2 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 2 | 4 | 5 | 6 | 2 | 5 | 2 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 5 | 3 | 6 | 4 | 0 | 4 | 0 | 2
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0
Stoma site pruritus (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 2 | 4 | 6 | 5 | 2 | 1 | 2 | 1
Amylase increased (Investigations) | 0 | 5 | 1 | 6 | 5 | 0 | 2 | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 6 | 2 | 4 | 7 | 3 | 3 | 2 | 2
Blood alkaline phosphatase increased (Investigations) | 0 | 4 | 4 | 4 | 4 | 2 | 3 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1 | 4 | 8 | 11 | 1 | 7 | 0 | 3
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 2 | 4 | 3 | 1 | 1 | 0 | 0
Lipase increased (Investigations) | 0 | 4 | 1 | 6 | 5 | 1 | 4 | 1 | 3
Lymphocyte count decreased (Investigations) | 0 | 4 | 1 | 4 | 3 | 1 | 3 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0 | 4 | 0 | 0
Platelet count decreased (Investigations) | 0 | 5 | 2 | 1 | 2 | 0 | 4 | 0 | 1
Weight decreased (Investigations) | 0 | 5 | 9 | 3 | 11 | 2 | 6 | 0 | 2
White blood cell count decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 15 | 29 | 17 | 14 | 15 | 20 | 3 | 7
Dehydration (Metabolism and nutrition disorders) | 1 | 3 | 6 | 5 | 8 | 1 | 4 | 0 | 3
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 1 | 1 | 2 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 4 | 3 | 4 | 6 | 0 | 4 | 0 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 3 | 3 | 1 | 2 | 0 | 1 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 3 | 4 | 2 | 4 | 2 | 2 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2 | 6 | 2 | 7 | 3 | 3 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 4 | 5 | 6 | 10 | 2 | 4 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 4 | 3 | 2 | 2 | 2 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 11 | 10 | 20 | 11 | 10 | 9 | 3 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 9 | 3 | 11 | 8 | 10 | 16 | 1 | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2 | 0 | 2 | 8 | 1 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3 | 1 | 1 | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 3 | 4 | 3 | 1 | 1 | 6 | 0 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 2 | 6 | 1 | 7 | 0 | 5 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 4 | 3 | 6 | 3 | 3 | 9 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 5 | 0 | 3 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 6 | 4 | 11 | 8 | 0 | 3 | 0 | 1
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 9 | 7 | 6 | 5 | 4 | 8 | 2 | 3
Dysgeusia (Nervous system disorders) | 0 | 1 | 1 | 2 | 3 | 1 | 5 | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 5 | 1 | 7 | 4 | 4 | 7 | 0 | 2
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 2 | 2 | 0 | 1 | 0 | 7 | 0 | 1
Polyneuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 2 | 1 | 0 | 2 | 1 | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 1 | 0
Agitation (Psychiatric disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 5 | 0 | 5 | 1 | 2 | 3 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 1
Depression (Psychiatric disorders) | 0 | 1 | 3 | 3 | 0 | 0 | 2 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 2 | 5 | 6 | 4 | 2 | 9 | 0 | 2
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 3 | 3 | 3 | 1 | 3 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 4 | 1 | 0 | 2 | 1 | 1 | 1
Haematuria (Renal and urinary disorders) | 0 | 3 | 3 | 4 | 3 | 3 | 13 | 1 | 2
Nocturia (Renal and urinary disorders) | 0 | 1 | 3 | 1 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 4 | 2 | 1 | 2 | 1 | 3 | 1 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 1 | 2 | 1 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 1 | 4 | 3 | 0 | 3 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 3 | 2 | 1 | 1 | 2 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 13 | 8 | 7 | 6 | 2 | 6 | 1 | 3
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 9 | 7 | 6 | 6 | 7 | 10 | 2 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 2 | 1 | 1 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Nasal septum perforation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 2 | 1 | 0 | 1 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 2 | 0 | 4 | 1 | 2 | 1 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 1 | 1 | 4 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 3 | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 2 | 3 | 2 | 4 | 1 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 12 | 6 | 13 | 10 | 10 | 7 | 2 | 5
Rash (Skin and subcutaneous tissue disorders) | 0 | 9 | 7 | 10 | 7 | 6 | 6 | 0 | 5
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 11 | 10 | 8 | 5 | 2 | 4 | 1 | 4
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 2 | 1 | 1 | 0 | 1 | 0
Flushing (Vascular disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 1 | 2 | 3 | 2 | 1 | 0 | 4 | 0 | 1
Hypertension (Vascular disorders) | 0 | 4 | 1 | 4 | 3 | 1 | 2 | 0 | 1
Hypotension (Vascular disorders) | 0 | 2 | 4 | 3 | 4 | 2 | 2 | 1 | 1
Superficial vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-01): https://cdn.clinicaltrials.gov/large-docs/57/NCT02985957/Prot_SAP_000.pdf